CLINICAL TRIAL: NCT02161094
Title: Diabetes Incentive Performance Study（DIPS）at Shanghai Jiading District
Brief Title: Diabetes Incentive Performance Study (DIPS) at Shanghai Jiading District
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCEMD-019
Record Dates: First submitted 2014-05-25; First posted 2014-06-11 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: Community management incentives
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Physicians (Experimental): Give incentives to physicians based on their patient's HbA1c improvement
  Interventions: Behavioral: Give incentives to patients based on their own HbA1c improvement
- Group 2: Diabetic patients (Experimental): Give incentives to patients based on their own HbA1c improvement
  Interventions: Behavioral: Give incentives to physicians based on their patient's HbA1c improvement
- Group 3: Both Physicians and Patients (Experimental): Give incentives to both based on the HbA1c improvements from the physicians' patients
  Interventions: Behavioral: Give incentives to physicians based on their patient's HbA1c improvement; Behavioral: Give incentives to patients based on their own HbA1c improvement
- Group 4: Control group (No Intervention): Receive no incentive but will be provided diabetes education booklet and group education courses for DM control as usual

INTERVENTIONS:
Behavioral: Give incentives to physicians based on their patient's HbA1c improvement
  Arms: Group 2: Diabetic patients; Group 3: Both Physicians and Patients
Behavioral: Give incentives to patients based on their own HbA1c improvement
  Arms: Group 1: Physicians; Group 3: Both Physicians and Patients

SUMMARY:
Objectives:Physicians from the Shanghai Jiading community clinic were invited to attend the study seminar. Those physicians who meet the criteria of the study plan were being selected to participate voluntarily. From their patient's record, the physicians will recruit a total of 1300 patients with type 2 diabetes who meet the criteria of the Jiading Study.

The study utilizes the social learning theory that motivation and social support are important to make behavioral change. The mechanism of providing incentive for patients and physicians will be established after the permission from the Internal Review Board of the hospital and will be approved by the hospital director. Physicians and their patients were randomly divided into 4 groups: Group 1- Physicians only; Group 2 - Patients only; Group 3 - Both Physicians and Patients, Group 4 - control. Groups 1-3 will receive incentives if they can maintain the ideal level of Hemoglobin A1c (HbA1c) during the 3-years study period. The forth group serves as a control and will not receive any incentive but will be provided diabetes education booklet and group education courses for DM control as usual. Based on the annual evaluation of the level of improvement on HbA1c that is a joint effort of both patients and physicians to achieve the targeted goal of adequate HBA1c level, the value of incentives will be increased accordingly. Our ultimate goal is to evaluate the effectiveness of incentive as an intervention tool to improve the health status of the diabetic patients.

DETAILED DESCRIPTION:
Methods：

This study is an open- label controlled randomized cluster trial and will invite eligible physicians and their patients to attend the study. These physicians work in health community center at Shanghai Jiading district and their patients are from the district community. Each physician should care and monitor at least 20 of his or her patients. This serves as a cluster randomized unit. The study size consists of 40 or more units within the Jiading District of Shanghai. Samples will taken from these patients according to the preset schedule and will measure patients' level of HbA1c accordingly. The physicians will recruit their patients who meet the criterion of the Jiading Study Standard. All of these patients have established their own health record by physicians in the community health center. To the enrolled patients, the study will obtain the information such as demographic characteristics, diagnosis and treatment, complications , various of biochemical index, skill and capacity of disease self-management, etc. Biomarkers and genetic risk factors will be evaluated in the study subjects. The study also will give several training courses to the enrolled physicians and the patients, all of them need to meet the study criteria and will sign the inform consent to participate in the study.

The study will use the method of randomized complete block design to classify the enrolled units into 4 groups. Group 1- Physicians only; Group 2 - Patients only; Group 3 - Both Physicians and Patients, Group 4 - control. Groups 1-3 will receive incentives if they can obtain or/and maintain the ideal level of Hemoglobin A1c (HbA1c) during the 3-years study period. We aim to achieve a target of HbA1c < 7% or to reduce 0.5% HbA1c level annually during 3 years study period. The incentive is in the form of cash or same value awards. The amount of the incentives will increase annually depending upon the change of HbA1c. The award is served as an motivation factor and token for rewarding the desire for self-discipline and disease management to enhance self-efficacy. The control group will not receive any incentives but will be provided diabetes education booklet and group education courses for DM control as usual.

The study will use the existing tele-medicine system to monitor patients' blood pressure and blood glucose remotely. The system of the telemedicine will also provide a series of diabetes education and training courses to support the physicians and the patients about the diabetes treatment, care and the self-management on the diseases. The study will document the changes on the patients' blood pressure, biochemical index, medication, quality of life, self-management skill of diabetes, life behavior, complications and costs.

Endpoint of the study:

The study will be ended in 36 months, endpoint measurement indicators are listed below:

1. Withdraw rate: Patient who drop out from the study;
2. Diabetic complication rate: Patient with new complications, such as macro- or micro-vascular complications;
3. Admission rate due to diabetic related illness： Patient's diabetic condition worsen, needs to be hospitalized or surgery;
4. Frequency of hypoglycemia incidences：Patient who has frequently severe hypoglycemia or other complications that can not continue the study;
5. Mortality rate among enrolled patients Death.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed type 2 diabetes patients (ICD9) according to the medical record and patient's disease history；
2. Diagnosis type 2 diabetes more than 6 months;
3. Receive DM therapy and follow up in health community center for more than 12 years;
4. Are insured for social health insurance system for treatment and medication reimbursement;
5. agree to participate in the study and have signed the Inform Consent Form.

Exclusion Criteria:

1. Terminal illness；
2. Hearing loss or severe visual disorder;
3. Planned to receive selective surgery within 3months;
4. Are in Pregnancy or breast-feeding while study;
5. Observed mental confusion suggesting dementia;
6. Ongoing psychiatric care;
7. Paralysis or residence in a long-term care facility;
8. Life expectancy is less than 12 months.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 36months

SECONDARY OUTCOMES:
Fasting plasma glucose FPG | 36months
Fast serum insulin FINS | 36months
Metabolic parameters | 36months
Serum lipids | 36months
Urine protein | 36months
BMI | 36months
Blood pressure | 36 months
Score on the Diabetes Quality Of Life | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD. PHD, Study Chair — Shanghai Clinical Centre for Endocrinology and Metabolism; Liebin Zhao, MSM, Study Chair — Center of Diabetes, Ruijin Hospital, Shanghai JiaoTong University School of Medicine; Yuhong Chen, MD, Study Chair — Shanghai Clinical Centre for Endocrinology and Metabolism, Ruijin Hospital, Shanghai JiaoTong University, School of Medicine
Locations (1):
- Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China